CLINICAL TRIAL: NCT07121478
Title: Lurbinectedin as a Second-line Treatment for High-grade Pancreatic Neuroendocrine Tumors
Brief Title: Patients With High-grade Pancreatic Neuroendocrine Tumors
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Seoul National Hospital (Other Government); Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sang Myung Woo, Principal investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2024-0187
Record Dates: First submitted 2025-06-15; First posted 2025-08-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Tumor of Pancreas; Pancreatic Neuroendocrine Tumors
Keywords: Lurbinectedin; Neuroendocrine Tumors
MeSH Terms: conditions — Adenoma, Islet Cell; Neuroendocrine Tumors | interventions — PM 01183; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Lurbinectedin shall be administered intravenously at a dose of 3.2 mg/m2 over 60 minutes every 21 days. The administration of the study drug shall be continued until disease progression or the occurrence of unacceptable toxicity.
  Interventions: Drug: Lurbinectedin 4 MG Injection [Zepzelca]

INTERVENTIONS:
Drug: Lurbinectedin 4 MG Injection [Zepzelca] — Lurbinectedin shall be administered intravenously at a dose of 3.2 mg/m2 over 60 minutes every 21 days. The administration of the study drug shall be continued until disease progression or the occurrence of unacceptable toxicity.

SUMMARY:
* Pancreatic neuroendocrine tumor (pNET) is a rare form of cancer. Treatment options such as hormonal therapy (octreotide) and targeted therapy (everolimus and sunitinib) may be considered for grade 1 or 2 pNETs; however, cytotoxic chemotherapy is essential in cases with grade 3 pNETs or pNECs.
* Cisplatin/etoposide remains the treatment of choice for high-grade pNET/pNEC. Other irinotecan-based therapies, such as FOLFIRI (cisplatin/irinotecan), FOLFOX, and temozolomide ± capecitabine, have been employed; however, a standard of care remains to be established.

DETAILED DESCRIPTION:
* Lurbinectedin, a selective inhibitor of oncogenic transcription, recently received accelerated FDA approval for lung cancer (small cell type) after demonstrating efficacy in an open-label, phase II basket study (ORR 35%, mOS 9.3 months, mPFS 3.5 months).
* A previous study that involved patients with grade 2 or higher NET/NEC who had undergone treatment with lurbinectedin revealed that the ORR, mOS, and mPFS of the six patients with pNET was 6.5%, 7.4 months, and 1.4 months, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Pancreatic neuroendocrine tumor or neuroendocrine carcinoma
* Documented failure of prior standard anti-cancer treatment
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm³
* Platelet count ≥ 100,000 cells/mm³
* Ability to understand study content, willingness to comply with study procedures, and commitment to complete the study

Exclusion Criteria:

* Currently receiving treatment for other cancers (except those who completed treatment and have been disease-free for at least 2 years prior to enrollment)
* Pregnant or breastfeeding women
* Deemed unsuitable for participation by the investigator due to clinical or medical reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The overall response rate | From date of first administration of drug until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24months"
  The proportion of participants who achieve a complete response (CR) or partial response (PR) as determined by the investigators according to the Response Evaluation Criteria in Solid Tumors

SECONDARY OUTCOMES:
Disease control rate | From date of the first administration of drug until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  1. Disease control is defined as the proportion of participants achieving complete response (CR), partial response (PR), or stable disease (SD) as assessed by investigators per RECIST v1.1 criteria.
Duration of response | From date of first documented response until the date of disease progression, relapse, or death from any cause, whichever occurs first, assessed up to 24 months.
  from date of first response to the date of disease progression, relapse, or death
Progression-free survival | From the date of first infusion until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
  time from the date of first infusion to disease progression or death from any cause
Overall survival | from the date of first infusion until death from any cause or loss to follow-up, whichever occurs first, assessed up to 24 months.
  from the date of first infusion to death or loss to follow-up
Evaluate the safety and tolerability of Lurbinectedin | From the date of first infusion until disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

OTHER OUTCOMES:
Tissue and blood sampling for discovering biomarkers | Every 6 weeks (two 28-day cycles) until the end of Cycle 6, and then every 9 weeks (three 28-day cycles) until documented disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
  Biomarker should be identified by statistical methods for correlation between disease control rates, response duration, progression-free survival, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Myung Woo(Principal), MD, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Plans for sharing individual participant data have not yet been finalized.

REFERENCES:
- [Background] Zhang MY, He D, Zhang S. Pancreatic neuroendocrine tumors G3 and pancreatic neuroendocrine carcinomas: Differences in basic biology and treatment. World J Gastrointest Oncol. 2020 Jul 15;12(7):705-718. doi: 10.4251/wjgo.v12.i7.705. PMID 32864039
- [Background] Trigo J, Subbiah V, Besse B, Moreno V, Lopez R, Sala MA, Peters S, Ponce S, Fernandez C, Alfaro V, Gomez J, Kahatt C, Zeaiter A, Zaman K, Boni V, Arrondeau J, Martinez M, Delord JP, Awada A, Kristeleit R, Olmedo ME, Wannesson L, Valdivia J, Rubio MJ, Anton A, Sarantopoulos J, Chawla SP, Mosquera-Martinez J, D'Arcangelo M, Santoro A, Villalobos VM, Sands J, Paz-Ares L. Lurbinectedin as second-line treatment for patients with small-cell lung cancer: a single-arm, open-label, phase 2 basket trial. Lancet Oncol. 2020 May;21(5):645-654. doi: 10.1016/S1470-2045(20)30068-1. Epub 2020 Mar 27. PMID 32224306
- [Background] Longo-Munoz F, Castellano D, Alexandre J, Chawla SP, Fernandez C, Kahatt C, Alfaro V, Siguero M, Zeaiter A, Moreno V, Sanz-Garcia E, Awada A, Santaballa A, Subbiah V. Lurbinectedin in patients with pretreated neuroendocrine tumours: Results from a phase II basket study. Eur J Cancer. 2022 Sep;172:340-348. doi: 10.1016/j.ejca.2022.06.024. Epub 2022 Jul 10. PMID 35830841